CLINICAL TRIAL: NCT01036802
Title: An Exploratory Study of Anticoagulation For Pulmonary Hypertension in Sickle Cell Disease
Brief Title: Anticoagulation For Pulmonary Hypertension in Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in accruing subjects
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-1596; R01HL094592-01A1 (NIH)
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Hypertension
Keywords: sickle cell disease; pulmonary hypertension; coagulation activation; platelet activation; endothelial activation
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warfarin (Active Comparator): Patients on the active treatment arm will be anticoagulated using the vitamin K antagonist, warfarin
  Interventions: Drug: Warfarin
- Placebo (Placebo Comparator): matching active products
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Warfarin — Patients on the active treatment arm will receive warfarin to achieve a target international normalized ratio of between 2 and 3
  Other Names: Coumadin
  Arms: Warfarin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Sickle cell disease (SCD) is often referred to as a hypercoagulable state. However, the contribution of coagulation activation to the pathogenesis of SCD remains uncertain. Pulmonary hypertension (PHT) is a common complication associated with significant morbidity and mortality. Autopsy studies of SCD patients with PHT show evidence of in situ thrombosis involving pulmonary vessels, similar to findings in non-sickle cell patients with PHT. Anticoagulation has been reported to be of benefit in non-sickle cell patients with PHT. With the evidence of increased coagulation activation in SCD, PHT represents a clinical endpoint that may be used to evaluate the contribution of coagulation activation to the pathophysiology of SCD. The investigators hypothesize that increased thrombin generation, as well as platelet activation are central to the pathophysiology of SCD and contribute to the occurrence of several SCD-related complications, including PHT. As a consequence, treatment modalities that down-regulate thrombin generation would be expected to delay the progression of PHT and result in improved survival in patients with SCD.

DETAILED DESCRIPTION:
As a result of the presence of large vessel thrombotic complications, as well as the biochemical evidence of ongoing coagulation activation, sickle cell disease (SCD) is often referred to as a hypercoagulable state. However, the contribution of coagulation activation to the pathogenesis of SCD remains uncertain. While the majority of clinical studies using anticoagulants have shown no convincing benefit in the prevention or treatment of acute pain episodes, most of these studies were small and poorly controlled. Furthermore, because the acute pain episode appears to result from the occlusion of postcapillary venules by the interaction of red blood cells and other cellular elements with the vascular endothelium and subendothelial matrix proteins, it may not be the ideal clinical endpoint for assessing the effect of anticoagulation in SCD patients. Pulmonary hypertension (PHT), a common complication associated with significant morbidity and mortality, and with histopathologic findings of in situ thrombosis involving pulmonary vessels, represents a clinical endpoint that is likely due, at least in part, to increased thrombin generation, and may therefore be used to evaluate the contribution of coagulation activation to the pathophysiology of SCD. Twenty patients with sickle cell anemia (HbSS) or sickle beta zero thalassemia (Sickle beta zero thalassemia) and mild PHT who meet the eligibility requirements will be enrolled, 10 patients to receive anticoagulation with warfarin and 10 to receive placebo rfor 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years of age
* Have a confirmed diagnosis of sickle cell anemia (HbSS) or sickle cell beta zero thalassemia
* Have evidence of persistent elevation of pulmonary artery systolic pressure on Doppler echocardiography (TR jet velocity of 2.5 to 2.9 m/s [or estimated pulmonary artery systolic pressure above the upper limit of reference adjusted ranges and up to 45 mm Hg]), but no evidence of moderate or severe diastolic dysfunction on tissue Doppler echocardiography. Mild PHT must be confirmed on repeat evaluation, at least 3 months later
* Have a serum creatinine =/< 1.5 mg/dl
* Have serum transaminase values (ALT) < 2 times upper limits of normal
* Have serum albumin =/> 3.2 g/dl
* Have a platelet count =/< 150,000 cu/mm
* Have normal baseline coagulation profile (PT/PTT)
* Patients on treatment with hydroxyurea should be on a stable dose for at least 6 months. Doses of hydroxyurea may only be adjusted during the course of the study for safety reasons.
* Be able to understand the requirements of the study and be willing to give informed consent.
* Women of childbearing age must be practicing (and will continue to practice for the course of the study) an adequate method of contraception.

Exclusion Criteria:

* Have a baseline hemoglobin < 6.0 gm/dl
* Have congenital heart disease, valvular heart disease, and other identified cause of pulmonary hypertension (including pulmonary fibrosis) unrelated to SCD
* Have an elevated pulmonary capillary wedge pressure, as evidenced by E/Em > 15 by pulsed wave and tissue Doppler imaging
* Have no measurable tricuspid regurgitant velocity on echocardiography
* Have a history of major gastrointestinal bleeding or a bleeding diathesis
* Have sickle cell complications such as recent vaso-occlusive crisis or acute chest syndrome, 4-weeks prior to commencing the study
* Have a history of clinically overt stroke(s) or seizures
* Have a brain magnetic resonance imaging/magnetic resonance angiography scan with evidence of Moya Moya within the preceding year
* Are pregnant or breastfeeding
* Are on chronic anticoagulant therapy
* Have a history of metastatic cancer
* Are chronically on therapy with aspirin or non-steroidal anti-inflammatory agents
* Are on a chronic transfusion program or have received a blood transfusion in the prior 8 weeks
* Have a positive urine toxicology screen for cocaine and amphetamines
* Have a history of alcohol abuse
* Are currently receiving treatment with epoprostenol (or similar prostacyclin analog), sildenafil (or similar phosphodiesterase 5 inhibitor), bosentan or arginine
* Have ingested any investigational drugs within the past 4 weeks.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized 1:1 to receive anticoagulation with warfarin or placebo after evaluation in the clinical and translational research center. Enrollment began in January 2010 and ended in September 2012 due to poor patient accrual.
Pre-assignment Details: Following patient identification, an open-label run-in period was begun to ensure patient doses of warfarin could be titrated to a stable level that achieved an international normalized ratio between 2.0 and 3.0 without exceeding a dose of 15 mg per day and to exclude patients with a level of compliance less than 80% (based on pill counts).
Groups:
- Placebo: Patients were randomized to placebo
Period: Overall Study
Arm/Group | Warfarin | Placebo
Started | 2 | 1
Completed | 2 | 1 (Patient was taken off study after 7 months as she required hip replacement surgery.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (12.02) | 53 | 37.3 (16.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of Anticoagulation on Pulmonary Artery Systolic Pressure Was Obtained by Doppler Echocardiography
Description: We determined the effect of anticoagulation with warfarin on estimated pulmonary artery systolic pressure obtained by Doppler echocardiography. The presented data are average values for the study subjects in the treatment group. When data was missing, the previous value was carried forward.
Time Frame: Measurements were obtained at Screening, and at Months 3, 6, 9, and 12
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 2 | 1
mm Hg
  Screening (n=2,1) | 41.3 (0) [39 to 43.6] | 43.6 (0) [43.6 to 43.6]
  Month 3 (n=1,1) | 39.2 [39.2 to 39.2] | 39.2 [39.2 to 39.2]
  Month 6 (n=2,1) | 41.3 [39.2 to 43.6] | 43.6 [43.6 to 43.6]
  Month 9 (n=1,1) | 46 [46 to 46] | 37 [37 to 37]
  Month 12 (n=1,1) | 46 [46 to 46] | 37 [37 to 37]

2. Secondary Outcome: 6-minute Walk Test
Description: We evaluated the distance walked over 6 minutes. The presented data are average values for the study subjects in the treatment group. When data was missing, the previous value was carried forward.
Time Frame: Measurements were obtained at Screening, Months 3, 6, 9, and 12
Measure: Mean (Full Range); unit: feet
Groups:
- Placebo: Patients were on placebo
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 2 | 1
feet
  Screen (n=1,1) | 1381 (0) [1381 to 1381] | 1135 (0) [1135 to 1135]
  Month 3 (n=1,1) | 1275 [1275 to 1275] | 1135 [1135 to 1135]
  Month 6 (n=1,1) | 1275 [1275 to 1275] | 1075 [1075 to 1075]
  Month 9 (n=1,1) | 1275 [1275 to 1275] | 1075 [1075 to 1075]
  Month 12 (n=1,1) | 1275 [1275 to 1275] | 1075 [1075 to 1075]

3. Secondary Outcome: Thrombin Generation
Description: We evaluated the effect of warfarin on a plasma measure of thrombin generation (thrombin-antithrombin complex)
Time Frame: Measurements were obtained at Screening, and at Months 3, 6, 9, and 12
Population: No analysis was performed due to the early termination of the study and the very small number of participating subjects.
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Platelet Activation
Description: We evaluated the effect of anticoagulation with warfarin on platelet activation assessed by measuring plasma levels of soluble CD40 ligand
Time Frame: Measurements were obtained at Screening, Prior to Run-in, and at Months 3, 6, 9, and 12
Population: No analysis was performed due to the early termination of the study and the very small number of participating subjects.
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Endothelial Activation
Description: We assessed the effect of warfarin on plasma measures of endothelial activation (soluble vascular cell adhesion molecule-1)
Time Frame: Measurements were obtained at Screening, and at Months 3, 6, 9, and 12
Population: As the number of subjects studied were very few, requiring discontinuation of the study, evaluation of endothelial activation was not performed.
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: All-cause Mortality
Description: We assessed the effect of warfarin on mortality in the study subjects
Time Frame: Assessment was obtained until completion of study at 12 months
Measure: Number; unit: participants
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 2 | 1
participants | 0 | 0

7. Secondary Outcome: Major and Minor Bleeding Complications
Description: We evaluated the safety of warfarin by evaluating for major and minor bleeding complications in study subjects
Time Frame: Evaluations were obtained at Screening, and at Months 3, 6, 9, and 12
Measure: Number; unit: participants
Arm/Group | Warfarin | Placebo
Number analyzed (Participants) | 2 | 1
participants
  Screen | 0 | 0
  Month 3 | 0 | 0
  Month 6 | 0 | 0
  Month 9 | 0 | 0
  Month 12 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Warfarin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin (N=2) | Placebo (N=1)
Delayed hemolytic transfusion reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Subject was transfused following hospitalization for a pain crisis, but was readmitted 1 week following discharge with findings consistent with a delayed hemolytic transfusion reaction.

LIMITATIONS AND CAVEATS:
This study was terminated early due to difficulty in accruing subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No